CLINICAL TRIAL: NCT04306614
Title: Capillary Versus Suction Needle Aspiration for Rapid Onsite Cytologic Evaluation in Endobronchial Ultrasound Biopsies
Brief Title: Capillary Versus Suction Needle Aspiration for Endobronchial Ultrasound (EBUS) Biopsies.
Acronym: CAPSUNN-EBUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 1
Record Dates: First submitted 2020-03-03; First posted 2020-03-13 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2020-02

CONDITIONS: Lung Cancer; Mediastinal Lymphadenopathy; Thoracic Cancer
Keywords: Endobronchial Ultrasound; Rapid-Onsite Cytologic Evaluation; Procedure duration
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capillary technique (Experimental)
  Interventions: Procedure: Endobronchial Ultrasound guided Transbronchial Fine Needle Aspiration
- Suction technique (Placebo Comparator)
  Interventions: Procedure: Endobronchial Ultrasound guided Transbronchial Fine Needle Aspiration

INTERVENTIONS:
Procedure: Endobronchial Ultrasound guided Transbronchial Fine Needle Aspiration — Bronchoscopic procedure to allow for sampling mediastinal lymphadenopathy or proximal lung tumours under real-time ultrasound guidance.

SUMMARY:
Endobronchial ultrasound (EBUS)-guided transbronchial needle aspiration is a procedure used to obtain tissue samples (biopsies) of lymph nodes near the airways or of lung tumours growing in close proximity to the airways. Briefly, an endoscope with an ultrasound probe which is inserted through the mouth and into the airways. Once in the airways, the ultrasound allows for identification of the optimal biopsy site; a hollow biopsy needle is then inserted into the tissue under real-time ultrasound visualization and a sample is extracted.

In the investigator's centre, the extracted sample is then immediately subjected to rapid on-site evaluation (ROSE). During the ROSE procedure, a cytotechnologist uses part of the sample to make a limited number direct smears which are then rapidly stained and evaluated under a microscope by the cytotechnologist. The cytotechnologist provides an assessment of the adequacy of the sample for diagnosis. The respirologist performing the EBUS then uses this information to: i) determine whether additional sampling is required, and ii) triage any additional samples for ancillary studies as needed. A final cytopathological diagnosis is established several days later, when all of the material from the procedure (including the material not evaluated at ROSE) is examined by a cytopathologist.

There are different techniques which are utilized to perform the needle aspiration biopsy. Suction aspiration (where pressure suction is applied to the needle to draw out material) which is the standard at many centres around the world and capilliary suction (where a tiny wire is drawn back slowly to create more gentle suction force) which is utilized often at LHSC.

The purpose of this study is to evaluate for differences in ROSE adequacy between these two methods.

ELIGIBILITY:
Inclusion Criteria:

* Patient age greater to or equal than 18 years old
* Receiving an endobronchial ultrasound for any diagnostic reason

Exclusion Criteria:

* Patients under 18 years old
* Patient refuses consent to undergo endobronchial ultrasound or is incapable of decision making.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Number of ROSE preparations per patient | During the procedure
Procedure Duration | During the procedure
Adequacy of ROSE sample (0-1) | During the procedure

SECONDARY OUTCOMES:
Adequate lymphocyte sampling (0-2) | During the procedure
Adequate diagnostic cells (0-2) | During the procedure
Amount of blood contamination on ROSE slide (0-2) | During the procedure
Adequacy of final specimen for ancillary testing (1-3) | During the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Inderdeep Dhaliwal, Principal Investigator — Assistant Professor
Locations (1):
- London Health Sciences Centre - Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No